CLINICAL TRIAL: NCT05966038
Title: ALS/MND Natural History Study Data Repository
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Henry Ford Health System (Other); Northwestern University (Other); Temple University (Other); St. Louis University (Other); University of Florida (Other); University of Minnesota (Other); Virginia Commonwealth University (Other); Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); Providence Health & Services (Other); University of Pittsburgh (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Lahey Clinic (Other); Hadassah Medical Organization (Other); Tel Aviv Medical Center (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Alexander Sherman, Director, Center for Innovation and Bioinformatics, Massachusetts General Hospital
Other Study IDs: 2013P001670; 5U01FD008125-02 (FDA); 2022A011556 (Other Grant/Funding Number: Biogen, Inc.); 2022A018800 (Other Grant/Funding Number: Mitsubishi Tanabe Pharma America)
Record Dates: First submitted 2023-06-15; First posted 2023-07-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: ALS; PLS; MND (Motor Neurone DIsease); Kennedy Disease; PMA - Progressive Muscular Atrophy; PBP - Progressive Bulbar Palsy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Bulbo-Spinal Atrophy, X-Linked; Muscular Atrophy, Spinal; Bulbar Palsy, Progressive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Participating sites may collect biofluids, including DNA, plasma, serum, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a data repository for multi-site multi-protocol clinic-based Natural History Study of ALS and Other Motor Neuron Disorders (MND).

All people living with ALS or other MNDs who attend clinics at the Study hospitals (sites) are offered to participate in the Study.

The Sites collect so-called Baseline information including demographics, disease history and diagnosis, family history, etc. At each visit, the Sites also collect multiple disease-specific outcome measures and events. The information is captured in NeuroBANK, a patient-centric clinical research platform.

The Sites have an option to choose to collect data into 20+ additional forms capturing biomarkers and outcome measures. Captured data after its curation are anonymized (all personal identifiers and dates are being removed), and the anonymized dataset is shared with medical researchers via a non-exclusive revocable license.

Funding Source - Biogen, Inc.; Mitsubishi Tanabe Pharma America; FDA OOPD.

DETAILED DESCRIPTION:
Most people with ALS or MND who are seen clinically by the PI or PI designees at participating sites will be recruited into this study. This well-established framework provides an opportunity to offer to a large proportion of people with ALS/MND a chance to participate in a clinical research project.

Upon obtaining consent, the following is done:

People with ALS/MND are assigned a Neurological Global Unique Identifier (NeuroGUID) and its study-specific derivative, NeuroSTAmP, which is used to link this Study's information to biological samples, images, and clinical data obtained from those individuals in this Study and other studies/trials, in which these patients participate(d).

The following information is captured in NeuroBANK platform:

Baseline information

* Longitudinal clinical and phenotypical data from routine clinical visits
* Longitudinal clinical and historical phenotypical data transcribed from electronic health records and notes
* Any other observational data that are of interest to the Investigator may be captured or linked to information in NeuroBANK.

Other Key Features

The site should track numbers of patients who declined participation. The site should have a mechanism in place to include an offer of participation to each patient in clinic (consenting does not require immediate data entry) Regular Data Quality checks may be performed at the site. Site personnel who intend to have access to NeuroBANK are trained and certified prior to given access.

Several registries, both cross-sectional and longitudinal, currently exist in ALS. NeuroBANK is distinct from other current registries in that it is a patient-centered platform that is designed to function as a data repository of patient data from clinical visits and multiple clinical research projects as well as linking these data to biorepository for tissue, imaging, and other biological information. This natural history study can act as a clinical research framework that may link clinical and clinical research data from current and past studies with biological specimens and image collections.

With obtained consents, biological specimens may be collected with bar-coded labels containing patient assigned study specific NeuroSTAmPs, printed from within NeuroBANK, and scanned into NeuroBANK's virtual distributed BioRepository module. Imaging studies are de-identified with NeuroSTAmPs and linked to clinical and phenotypical information. Anonymized clinical data obtained through this protocol are available to other researchers.

Study Population

Individuals who are seen during their clinical care visits are asked to allow their data to be uploaded and captured for clinical research. The NeuroBANK platform is located at and managed by the Center for Innovation and Bioinformatics (CIB), Neurological Clinical Research Institute (NCRI) of Massachusetts General Hospital (Boston, MA).

Consent Process

Every participant in the ALS clinic is approached to participate in this study. A signed informed consent form is obtained before any data are recorded for study purposes.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of El Escorial of suspected, possible, probable, or definite ALS or
* Other motor neuron disorders, including but not limited to Spinal-Bulbar Muscular Atrophy (SBMA, Kennedy's disease), Spinal Muscular Atrophy (SMA), Primary Lateral Sclerosis (PLS), Progressive Muscular Atrophy (PMA), and Progressive Bulbar Palsy (PBP)

Exclusion Criteria:

* Disease does not meet criteria for any motor neuron disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All people living with ALS/MND at participating multidisciplinary ALS/MND clinics
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | Every 3-4 months up to 5 years
  The ALS Functional Rating Scale revised is a 12-item rating scale that measures the progression of disability in patients with ALS. The ALSFRS-r assesses patients' levels of self-sufficiency in areas of feeding, grooming, ambulation and communication. The higher the score, the earlier in the disease progression.
  It consists of 12 questions with a maximum score of 48 points.
Slow Vital Capacity (SVC) | Every 3-4 months up to 5 years
  Slow vital capacity test normalized to age, sex, and height
Survival | Every 3-4 months up to 5 years
  Patient survival or survival equivalent (time to ventilator or feeding tube). Survival equivalent is assessed during routine clinical visits, while mortality event may be reported when becomes known to the treating clinician..

SECONDARY OUTCOMES:
Vital Signs | Every 3-4 months up to 5 years
  Vital Signs (Weight, BP, HR). Both systolic and diastolic pressure are measured.
Neurological Examination | Through study completion, annually up to 5 years
  Neurological exam that tests for abnormality various areas, from general assessment to coordination and cerebellar function, to sensation and reflexes, to cranial nerves and plantar
El Escorial Criteria | Through study completion, annually up to 5 years
  The El Escorial criteria are diagnostic criteria for ALS. They classify patients into categories of possible, probable, or definite ALS, based on signs of degeneration of upper and lower motor neurons in different body regions.
Handheld Dynamometry | Every 3-4 months up to 5 years
  Handheld Dynamometry for quantitative strength testing of 18 muscles that is a reliable and reproducible measure of decline in ALS
Grip Strength Testing | Every 3-4 months up to 5 years
  Grip Strength Testing
Rasch Overall ALS Disability Scale (ROADS) | Every 3-4 months up to 5 years
  Rasch Overall ALS Disability Scale, the ROADS provides a normed total score on 28 items from 0-146 to capture overall disability level in a linearly-weighted manner, with lower scores indicating disease progression
5 Times Sit to Stand | Every 3-4 months up to 5 years
  5 Times Sit to Stand Test
10 Meter Walk Test | Every 3-4 months up to 5 years
  10 Meter Walk Test
Physical Examination | Through study completion, annually up to 5 years
  Physical Examination that includes the following test areas for abnormality and clinical significance: respiratory, cardio, gastrointestinal, genitourinary. and musculoskeletal

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sherman, Principal Investigator — Massachusetts General Hospital
Locations (16):
- United States (12):
  - Loma Linda University Health, Loma Linda, California
  - Kaiser Permanente, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Providence ALS Clinic, Portland, Oregon
  - Temple University Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Tel Aviv Medical Center, Tel Aviv
- Italy (2):
  - Centro Clinico NEMO Milano, Milan
  - Istituti Clinici Scientifici Maugeri SpA, Milan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD are being shared with data requestors upon submission of the research proposal online. Data Access Committee reviews submissions and upon approval and execution of the Data Sharing Agreement, the dataset is provided to the data requestor.
Supporting Information: Study Protocol
Time Frame: 10-30 days from the initial request's online submission
Access Criteria: ALS/MND Natural History Consortium's Data Access committee reviews the merits of the requestors' research proposals and approves or denies data access

REFERENCES:
- See also: ALS/MND NATURAL HISTORY CONSORTIUM — https://www.data4cures.org/natural-history-consortium
- Available data/document: Individual Participant Data Set: NeuroGUID/NeuroSTAmP — https://www.data4cures.org/requestingdata — Anonymized data may be requested by submitting research proposal online. Data Access Committee will review the submission and upon its approval and execution of the Data Sharing Agreement, the dataset will be provided to the data requestor.